CLINICAL TRIAL: NCT01593085
Title: Evaluation of States in Major Depressive Patients With Cancer, Hospitalized in a Hospital Palliative
Acronym: DECAPAL
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: DECAPAL
Record Dates: First submitted 2012-04-30; First posted 2012-05-07 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2012-04

CONDITIONS: Cancer
Keywords: palliative cares; cancer; suicide risk
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients in palliative cares: patients with cancer in palliative cares An interview and will be offered to this patient during his hospitalization to be held (with the collection of personal and family psychiatric history of the patient, family and social context, the assessment of chronic pain and fatigue and quality of life,assessment of anxiety, Evaluation of symptoms of depression,asessment of suicide risk)
  Interventions: Behavioral: interview with a doctor for evaluating suicide risk

INTERVENTIONS:
Behavioral: interview with a doctor for evaluating suicide risk — patients with cancer in palliative cares An interview and will be offered to this patient during his hospitalization to be held (with the collection of personal and family psychiatric history of the patient, family and social context, the assessment of chronic pain and fatigue and quality of life,assessment of anxiety, Evaluation of symptoms of depression,asessment of suicide risk)
  --------------------------------------------------------------------------------

SUMMARY:
The investigators propose a study that aims to develop a methodology for assessing this risk and the psychological consequences of the malignancy in the palliative phase.

ELIGIBILITY:
Inclusion Criteria:

* Patient (s) age (s) 18 or more
* Patient (s) reach (s) of a cancer palliative stage
* Patient (s) hospital (s) in the palliative care service
* Patient (s) with cognitive function to an interrogation
* Patient (s) having a physical condition for an interview lasting 45 minutes
* Patient (s) that received clear information on the diagnosis and prognosis of their disease.
* Free and informed consent signed

Exclusion Criteria:

* Patient (s) age (s) under 18 years
* Patient (s) under supervision or unable to give informed consent
* Patient (s) whose cognitive functions do not allow an examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer in palliative cares
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
assessing the prevalence of suicide risk in patients with cancer admitted to a palliative care service. | at inclusion only, during hospitalization in palliative cares
  assessing the prevalence of suicide risk in patients with cancer admitted to a palliative care service.

SECONDARY OUTCOMES:
Evaluate the feasibility of a methodology for estimating the risk of suicide in patients with cancer admitted to a palliative care service | at inclusion only, during hospitalization in palliative cares
  Evaluate the feasibility of a methodology for estimating the risk of suicide in patients with cancer admitted to a palliative care service Questionnaires used are HADS Questionary, Scale HAMILTON, Scale BECK and Scale DUCHER
Assess the psychological impact of cancer pathology in patients in palliative | at inclusion only, during hospitalization in palliative cares
  Assess the psychological impact of cancer pathology in patients in palliative by evaluating depression score (with HADS HAMILTON, BECK, DUCHER scales)
Identify risk factors for suicide in this patient population | at inclusion only, during hospitalization in palliative cares
  Identify risk factors for suicide in this patient population with evaluation of type of cancer, psychiatric history, family and social context, quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine GRACH, MD, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre François BACLESSE, Caen, Calvados, France